CLINICAL TRIAL: NCT03286543
Title: A Prospective, Comparative Effectiveness Randomized Controlled Trial of SPR Peripheral Nerve Stimulation (PNS) Therapy for the Treatment of Pain Following Total Knee Arthroplasty (TKA) Utilizing Preoperative Lead Placement
Brief Title: Electrical Stimulation for the Treatment of Pain Following Total Knee Arthroplasty Using the SPRINT Beta System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0144-CSP-000
Record Dates: First submitted 2017-08-31; First posted 2017-09-18 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Total Knee Replacement; Total Knee Arthroplasty; Pain; Postoperative Pain; Orthopedic Disorder
Keywords: electrical stimulation; neurostimulation; TKA pain; pain following total knee replacement; total knee arthroplasty
MeSH Terms: conditions — Pain; Pain, Postoperative; Musculoskeletal Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Half of the subjects enrolled will be randomized (like flipping a coin) to the treatment group and half will be randomized to the control group. Both groups will receive the standard of care for pain management following total knee replacement surgery. Subjects in the treatment group will receive SPR's SPRINT Beta Peripheral Nerve Stimulation (PNS) System in addition to standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group (SPRINT Beta System) (Experimental): Subjects in the treatment group will have up to 2 leads placed in their leg that underwent total knee replacement, will use the SPRINT Beta System, and will receive electrical stimulation in addition to the standard of care.
  Interventions: Device: SPRINT Beta System
- Control Group (No Intervention): Subjects in the control group will receive the standard of care.

INTERVENTIONS:
Device: SPRINT Beta System — The SPRINT Beta System is an Investigational Device which delivers mild electrical stimulation to nerves in the leg that underwent lead placement. The SPRINT Beta System includes a small wire (called a "Lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Beta Stimulator).
  Other Names: SPRINT Beta Peripheral Nerve Stimulation (PNS) System; SPRINT Peripheral Nerve Stimulation (PNS) System; SPRINT System
  Arms: Treatment Group (SPRINT Beta System)

SUMMARY:
The purpose of this study is to determine if electrical stimulation (small levels of electricity) in addition to the standard of care can safely and effectively reduce pain following total knee replacement more than the standard of care, alone. This study involves a device called the SPRINT Beta System. The SPRINT Beta System delivers mild electrical stimulation to nerves in the leg that received the knee replacement. The SPRINT Beta System includes a small wire (called a "lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Beta Stimulator). About half the subjects in this study will receive the SPRINT Beta system (treatment group) and half will not (control group). Both groups will receive the standard of care.

ELIGIBILITY:
Key Inclusion Criteria:

* Scheduled to undergo a primary unilateral total knee replacement procedure

Key Exclusion Criteria:

* Body Mass Index > 40 kg/m2
* Conditions that place the subject at increased risk of infection
* History of valvular heart disease
* Implanted electronic device
* Bleeding disorder
* Allergy to skin surface electrodes and/or medical-grade adhesive tapes
* Pregnant

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California San Diego, La Jolla, California
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Joint Implant Surgeons, New Albany, Ohio
  - HD Research, Bellaire, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2017 (with first subject enrollment in September 2017) and was concluded in February 2020. Subjects were screened from the available pool of candidates scheduled to undergo a primary unilateral total knee replacement procedure.
Pre-assignment Details: After obtaining informed consent, subjects were evaluated for eligibility.
Groups:
- Consented Subjects: Subjects who signed an informed consent form.
- Treatment Group: Subjects in the Treatment Group were consented, scheduled to undergo a unilateral total knee arthroplasty (TKA), and met all eligibility criteria prior to randomization. These subjects had at least one Lead placed in their affected leg prior to TKA and used the SPRINT Beta System to receive electrical stimulation therapy in addition to the standard of care.
- Control Group: Subjects in the Control Group were consented, scheduled to undergo a unilateral total knee arthroplasty (TKA), and met all eligibility criteria prior to randomization. These subjects did not undergo Lead placement, and they received the standard of care following TKA.
Period: Consented
Arm/Group | Consented Subjects | Treatment Group | Control Group
Started | 47 | 0 | 0
Randomized (All subjects who were consented, met eligibility criteria, and were randomized.) | 45 | 0 | 0
Enrolled (Treatment Group subjects who were consented, randomized, and underwent Lead placement, AND Control Group subjects who were consented and randomized.) | 41 | 0 | 0
Intent to Treat Set (Subjects that were consented, randomized, enrolled, and progressed in study to designated randomization assignment therapy.) | 37 | 0 | 0
Per Protocol Set (Subjects that were consented, randomized, enrolled, have adequate diary completion, and continued study eligibility. Additionally, Treatment Group subjects must have received a Lead and experienced stimulation-evoked comfortable sensations or a reduction in pain with stimulation in the target area during Visit 2 (original or unscheduled) or Visit 4.) | 23 | 0 | 0
Completed | 28 | 0 | 0
Not Completed | 19 | 0 | 0
Not completed — Screen failure before randomization | 2 | 0 | 0
Not completed — Screen failure before enrollment | 4 | 0 | 0
Not completed — TKA cancelled after enrollment | 1 | 0 | 0
Not completed — Withdrawn from study | 12 | 0 | 0
Period: Study Enrollment
Arm/Group | Consented Subjects | Treatment Group | Control Group
Started | 0 | 18 | 23
Intent to Treat Set (Subjects that were consented, randomized, and enrolled.) | 0 | 18 | 19
Per Protocol Set (Subjects that were consented, randomized, enrolled, have adequate diary completion, and continued study eligibility. Additionally, Treatment Group subjects must have received a Lead and experienced stimulation-evoked comfortable sensations or a reduction in pain with stimulation in the target area during Visit 2 (original or unscheduled) or Visit 4.) | 0 | 7 | 16
Completed | 0 | 12 | 16
Not Completed | 0 | 6 | 7
Not completed — TKA cancelled after enrollment | 0 | 0 | 1
Not completed — Withdrawn from study | 0 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 18 | 23 | 41
Age, Categorical [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    number analyzed (Participants) | 18 | 22 | 40
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 11 | 20
    >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  years
    number analyzed (Participants) | 18 | 22 | 40
    (all) | 65.0 (5.5) | 63.0 (10.3) | 63.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    number analyzed (Participants) | 18 | 22 | 40
    Female | 12 | 12 | 24
    Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    number analyzed (Participants) | 18 | 22 | 40
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 18 | 21 | 39
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    number analyzed (Participants) | 18 | 22 | 40
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 16 | 21 | 37
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 23 | 41
Affected Leg [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    Right Leg: number analyzed (Participants) | 18 | 22 | 40
    Right Leg | 8 | 15 | 23
    Left Leg: number analyzed (Participants) | 18 | 22 | 40
    Left Leg | 10 | 7 | 17
Reason for Total Knee Arthroplasty (TKA) [Count of Participants; unit: Participants] — Population: One Control Group subject withdrew after randomization due to their unwillingness to participate as a control, and Demographic information was not collected.
  Participants
    Osteoarthritis: number analyzed (Participants) | 18 | 22 | 40
    Osteoarthritis | 16 | 21 | 37
    Post-Traumatic Arthritis: number analyzed (Participants) | 18 | 22 | 40
    Post-Traumatic Arthritis | 2 | 0 | 2
    Degenerative Joint Disease: number analyzed (Participants) | 18 | 22 | 40
    Degenerative Joint Disease | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Knee Pain While Walking
Description: All subjects were asked to complete daily diaries to record their average pain intensity while walking during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." For each subject, the mean score for each diary period was calculated and a mean of all four diary periods was calculated (weeks 1-4). The mean group scores for weeks 1-4 are reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA)
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
Scores on a scale | 3.70 (1.97) | 4.14 (1.49)

2. Primary Outcome: Number of Subjects That Experienced at Least One Study-Related Adverse Event
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition has occurred since their previous visit. If the subject experienced a change that was an adverse event, an Adverse Event Form was completed by the site. The number of Treatment Group subjects that experienced at least one study-related adverse event is reported here.
Time Frame: 30 months (from when the first Treatment Group subject enrolled to when the last Treatment Group subject completed the study)
Population: All enrolled Treatment Group subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
Participants | 8

3. Secondary Outcome: Average Knee Pain Over the Last 24 Hours
Description: All subjects were asked to complete daily diaries to track their average pain intensity during the past 24 hours over a 7-day period on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average score for each diary period was calculated across subjects, and the mean score for weeks 1-4 is reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA))
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
score on a scale | 3.24 (1.52) | 4.32 (1.34)

4. Secondary Outcome: Average Knee Pain at Rest
Description: All subjects were asked to complete daily diaries to track their average pain intensity at rest during the past 24 hours over a 7-day period on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average score for each diary period was calculated across subjects, and the mean score for weeks 1-4 is reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA))
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
score on a scale | 2.86 (1.23) | 3.48 (1.33)

5. Secondary Outcome: Pain Right Now as Measured by the Brief Pain Inventory
Description: Subjects were asked to rate their pain right now on an 11-point numerical scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The median score for each time point is reported. Baseline is considered Visit 2a (Lead Placement) for Treatment Group subjects and Visit 2b for Control Group subjects. For Treatment Group subjects for Visits 3, 4, 6, and 8, pain right now was assessed while peripheral nerve stimulation was on for at least one Lead. For Visit 4, the score reported during the last in-hospital day was used.
Time Frame: Baseline (Visit 2a/2b), Visit 3 (Day of Total Knee Arthroplasty (TKA)), Visit 4 (in-hospital), Visit 6 (2-weeks post TKA), and Visit 8 (4-weeks post TKA)
Population: Per Protocol Set - Data were not available for one Treatment Group subject at Visit 3 and for one Control Group subject at Visit 6.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
Scores on a scale
  Baseline | 1.0 [0 to 2] | 3.0 [1 to 10]
  Visit 3 (Day of TKA): number analyzed (Participants) | 6 | 16
  Visit 3 (Day of TKA) | 2.0 [0 to 8] | 2.0 [0 to 10]
  Visit 4 (In-Hospital) | 2.0 [1 to 6] | 3.5 [0 to 7]
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 6 (2-weeks Post-TKA) | 2.0 [1 to 8] | 3.0 [0 to 6]
  Visit 8 (4-weeks Post-TKA) | 1.0 [0 to 3] | 1.0 [0 to 6]

6. Secondary Outcome: Amount of Analgesic Usage
Description: Subjects recorded the amount/type of analgesics used in daily diaries. Narcotic usage was converted into morphine milligram equivalents (MME). Diaries were collected at various visits and were translated into post-operative days. The average MME was calculated for each subject for the first 28 days (4 weeks) following surgery, and the median of these averages across subjects was determined. If subjects had ceased opioid use (per the Recovery Milestones log), then missing scores following the date of opioid cessation were replaced with 0 MME. If diary entries were missing but the subject had not yet reported opioid cessation, then the missing value was replaced with the mean usage of the available days for the corresponding week. Subjects missing data from one or more entire diaries (i.e., weeks) and had not yet reported opioid cessation by the date of any missing diary were not included in this analysis.
Time Frame: Visits 5-8 (weeks 1-4 post-Total Knee Arthroplasty (TKA))
Population: Per Protocol Set - Data were not available for one Control Group subject at Visits 6-8.
Measure: Median (Full Range); unit: MME
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 14
MME
  Visit 5 (1-week Post-TKA) | 29.9 [3.2 to 49.3] | 31.4 [0.0 to 107.1]
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 6 (2-weeks Post-TKA) | 21.4 [2.1 to 31.1] | 22.5 [0.0 to 88.8]
  Visit 7 (3-weeks Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 7 (3-weeks Post-TKA) | 13.6 [1.1 to 20.0] | 17.1 [0.0 to 69.6]
  Visit 8 (4-weeks Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 8 (4-weeks Post-TKA) | 11.4 [0.0 to 20.7] | 2.9 [0.0 to 47.1]
  Average Across Visits 5-8: number analyzed (Participants) | 7 | 13
  Average Across Visits 5-8 | 19.1 [2.1 to 26.8] | 16.8 [0.13 to 75.0]

7. Secondary Outcome: Number of Subjects That Experienced at Least One Opioid-Related Side Effect
Description: Throughout the study, subjects were asked if they experienced any side effects related to opioid pain medications. The occurrences of these side effects were recorded and were not considered Adverse Events. The number of subjects that experienced at least one opioid-related side effect at each visit is reported. Baseline is considered Visit 2a (Lead Placement) for Treatment Group subjects and Visit 2b for Control Group subjects.
Time Frame: Baseline (Visit 2a/2b), Visits 4-11 (in-hospital days through 12-months post-Total Knee Arthroplasty (TKA))
Population: Per Protocol Set - Data were not available for one Treatment Group subject at Visit 6 and Visit 11.
  Data were not available for the following Control Group subjects: one at Visits 5, 6, 7, and 9, and three at Visits 10 and 11.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
Participants
  Baseline | 0 | 0
  Visit 4 (In-Hospital) | 3 | 7
  Visit 5 (1-week Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 5 (1-week Post-TKA) | 3 | 9
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 6 | 15
  Visit 6 (2-weeks Post-TKA) | 3 | 8
  Visit 7 (3-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 7 (3-weeks Post-TKA) | 2 | 6
  Visit 8 (4-weeks Post-TKA) | 1 | 4
  Visit 9 (2-months Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 9 (2-months Post-TKA) | 0 | 0
  Visit 10 (3-months Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 10 (3-months Post-TKA) | 0 | 0
  Visit 11 (12-months Post-TKA): number analyzed (Participants) | 6 | 13
  Visit 11 (12-months Post-TKA) | 0 | 0

8. Secondary Outcome: Timed Up and Go (TUG) Test
Description: Subjects began this test from a seated position in a standard chair and were timed while they stood up, walked to a marked point 10 feet away (at a normal, safe pace), returned to the chair, and sat down. Timed Up and Go (TUG) test times are expected to be greater immediately after surgery as compared to baseline.
Time Frame: Visit 1 (Baseline), Visit 4 (In-Hospital), Visit 6 (2-weeks Post-Total Knee Arthroplasty (TKA)), Visit 8 (4-weeks Post-TKA)
Population: Per Protocol Set - Data were not available for the following Control Group subjects: one at Visit 1 (subject was unable to complete test), three at Visit 4 (two subjects were unable to complete test), and one at Visit 6.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
seconds
  Time at Visit 1 (Baseline): number analyzed (Participants) | 7 | 15
  Time at Visit 1 (Baseline) | 12.44 [4.82 to 13.7] | 10.25 [7 to 26.24]
  Time at Visit 4 (In-Hospital): number analyzed (Participants) | 7 | 13
  Time at Visit 4 (In-Hospital) | 41.80 [11.13 to 141.32] | 42.22 [13.81 to 82.37]
  Time at Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Time at Visit 6 (2-weeks Post-TKA) | 14.28 [7.63 to 32.36] | 15.93 [7.39 to 56.0]
  Time at Visit 8 (4-weeks Post-TKA) | 10.68 [6.59 to 17.07] | 10.38 [6.9 to 40.68]

9. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The total distance that a subject could walk in 6 minutes was recorded, and subjects unable to walk at all were given a score of 0 meters. The median distance was then determined across subjects. 6 Minute Walk Test distances are expected to be reduced immediately after surgery as compared to baseline.
Time Frame: Visit 1 (Baseline), Visit 6 (2-weeks Post-Total Knee Arthroplasty (TKA)), Visit 8 (4-weeks post-TKA)
Population: Per Protocol Set - Data were not available for one Control Group subject at Visit 6.
Measure: Median (Full Range); unit: meters
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
meters
  Visit 1 (Baseline) | 458.5 [320.0 to 555.0] | 351.3 [0 to 504.0]
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 6 (2-weeks Post-TKA) | 280.0 [150.0 to 504.7] | 281.0 [0 to 680.2]
  Visit 8 (4-weeks Post-TKA) | 410.0 [270.0 to 693.0] | 329.0 [0 to 518.9]

10. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The Western Ontario McMaster University Osteoarthritis Index (WOMAC) questionnaire consists of 24 items that evaluate pain, stiffness, and physical functional disability. Each item is scored on an 11-point numerical rating scale from 0 to 10, where higher scores indicate greater pain, stiffness, and disability. For each subject, the scores from each of the 24 items were summed to calculate the subject's total score, with a minimum score of 0 and a maximum score of 240. The mean total score was then calculated across subjects for each time point.
Time Frame: Visit 1 (Baseline), Visit 3 (Day of Total Knee Arthroplasty (TKA)), Visit 6 (2-weeks post-TKA), Visit 8 (4-weeks post-TKA), Visit 10 (3-months post-TKA), and Visit 11 (12-months post-TKA)
Population: Per Protocol Set - Data were not available for one Treatment Group subject at Visit 11. Data were not available for the following Control Group subjects: three at Visit 3, one at Visit 6, three at Visit 10, and two at Visit 11.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
score on a scale
  Visit 1 (Baseline) | 87.00 (30.34) | 111.31 (38.78)
  Visit 3 (Day of TKA): number analyzed (Participants) | 7 | 13
  Visit 3 (Day of TKA) | 68.71 (47.87) | 99.23 (51.25)
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 6 (2-weeks Post-TKA) | 58.57 (33.24) | 81.13 (38.98)
  Visit 8 (4-weeks Post-TKA) | 40.29 (26.56) | 51.94 (30.83)
  Visit 10 (3-months Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 10 (3-months Post-TKA) | 22.86 (22.13) | 29.38 (21.05)
  Visit 11 (12-months Post-TKA): number analyzed (Participants) | 6 | 14
  Visit 11 (12-months Post-TKA) | 4.83 (4.36) | 12.79 (20)

11. Secondary Outcome: Number of Subjects Reporting Meaningful Improvement, Minimal or No Change, or Meaningful Worsening on the Patient Global Impression of Change (PGIC) Survey
Description: The Patient Global Impression of Change (PGIC) asks subjects to rate their improvement with treatment on a 7-point scale ranging from "very much worse" to "very much improved" as compared to before their knee replacement surgery. The subjects combine all the components of their experience into one overall score. Ratings of Much- or Very Much Improved are considered "Meaningful Improvements"; similarly, ratings of Much- or Very Much Worse are categorized as "Meaningfully Worse." Ratings of Minimally Improved, No Change, or Minimally Worse are considered "Minimal or No Change."
Time Frame: Visits 3-11 (Day of Total Knee Arthroplasty (TKA) through 12-months post-TKA)
Population: Per Protocol Set: Data were not available for one Treatment Group subject at Visit 11. Data were not available for the following Control Group subjects: one at Visit 4, one at Visit 6, one at Visit 9, three at Visit 10, and two at Visit 11.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
Participants
  Visit 3 (Day of TKA): Meaningful Improvement | 0 | 1
  Visit 3 (Day of TKA): Minimal or No Change | 5 | 14
  Visit 3 (Day of TKA): Meaningfully Worse | 2 | 1
  Visit 4 (In-Hospital): number analyzed (Participants) | 7 | 15
  Visit 4 (In-Hospital): Meaningful Improvement | 1 | 4
  Visit 4 (In-Hospital): Minimal or No Change | 5 | 9
  Visit 4 (In-Hospital): Meaningfully Worse | 1 | 2
  Visit 5 (1-week Post-TKA): Meaningful Improvement | 2 | 3
  Visit 5 (1-week Post-TKA): Minimal or No Change | 3 | 11
  Visit 5 (1-week Post-TKA): Meaningfully Worse | 2 | 2
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 6 (2-weeks Post-TKA): Meaningful Improvement | 2 | 3
  Visit 6 (2-weeks Post-TKA): Minimal or No Change | 3 | 11
  Visit 6 (2-weeks Post-TKA): Meaningfully Worse | 2 | 1
  Visit 7 (3-weeks Post-TKA): Meaningful Improvement | 2 | 3
  Visit 7 (3-weeks Post-TKA): Minimal or No Change | 3 | 12
  Visit 7 (3-weeks Post-TKA): Meaningfully Worse | 2 | 1
  Visit 8 (4-weeks Post-TKA): Meaningful Improvement | 2 | 6
  Visit 8 (4-weeks Post-TKA): Minimal or No Change | 3 | 9
  Visit 8 (4-weeks Post-TKA): Meaningfully Worse | 2 | 1
  Visit 9 (2-months Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 9 (2-months Post-TKA): Meaningful Improvement | 4 | 8
  Visit 9 (2-months Post-TKA): Minimal or No Change | 3 | 7
  Visit 9 (2-months Post-TKA): Meaningfully Worse | 0 | 0
  Visit 10 (3-months Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 10 (3-months Post-TKA): Meaningful Improvement | 6 | 9
  Visit 10 (3-months Post-TKA): Minimal or No Change | 1 | 4
  Visit 10 (3-months Post-TKA): Meaningfully Worse | 0 | 0
  Visit 11 (12-months Post-TKA): number analyzed (Participants) | 6 | 14
  Visit 11 (12-months Post-TKA): Meaningful Improvement | 6 | 12
  Visit 11 (12-months Post-TKA): Minimal or No Change | 0 | 2
  Visit 11 (12-months Post-TKA): Meaningfully Worse | 0 | 0

12. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) questionnaire has 13 questions that assess rumination, magnification, and helplessness. Subjects are asked to think back on painful experiences in the past and reflect on how often they had specific thoughts or feelings. Each of the 13 questions is scored on a 5-point scale where 0 represents "not at all," and 4 represents "all the time." The scores from each question were summed for each subject to provide a total PCS score, with a possible range from 0 to 52 with higher scores indicating a greater tendency to catastrophize pain (i.e. a higher score indicates a worse outcome). The median scores were then calculated across all subjects.
Time Frame: Visit 1 (Baseline), Visit 8 (4 weeks post-Total Knee Arthroplasty (TKA)), Visit 10 (3-months Post-TKA)
Population: Per Protocol Set - Data were not available for three Control Group subjects at Visit 10.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
score on a scale
  Visit 1 (Baseline) | 7 [0 to 13] | 7 [0 to 34]
  Visit 8 (4-weeks Post-TKA) | 6 [0 to 14] | 4 [0 to 19]
  Visit 10 (3-months Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 10 (3-months Post-TKA) | 1 [0 to 13] | 0 [0 to 15]

13. Secondary Outcome: Time to Meet Recovery Milestones up to Twelve Months Post-Total Knee Arthroplasty (TKA)
Description: Participants were queried at each visit from the date of their Total Knee Arthroplasty (TKA) until they met specific, post-surgical recovery milestones. Participants were queried up through the time at which they met each milestone or through their completion of the study, whichever came first (up to twelve months post-surgery). For each milestone, the median number of days between the date of TKA and date to achieve the milestone was calculated.
Time Frame: From Day of Surgery through completion of milestone or 12-months from Day of Surgery, whichever came first
Population: Per Protocol Set- Treatment Group: Data were not available for: 1 subject in "walked without assistive device", 1 in "cleared to drive". 1 subject did not cease opioids during the study. 5 subjects were retired and did not work.
  Control Group: Data were not collected for: 3 in "walked without assistive device", 2 in "able to climb stairs", 1 in "cleared to drive", 1 in "opioid cessation" (2 more did not cease opioids during the study). 9 subjects were retired and did not work.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
days
  Pain controlled without nerve block | 3 [1 to 5] | 2 [1 to 9]
  Walked with assistive device | 0 [0 to 1] | 1 [0 to 1]
  Walked without assistive device: number analyzed (Participants) | 6 | 13
  Walked without assistive device | 24 [2 to 52] | 16 [2 to 107]
  Walked 30 meters | 1 [0 to 16] | 4 [0 to 28]
  Able to climb flight of stairs: number analyzed (Participants) | 7 | 14
  Able to climb flight of stairs | 1 [0 to 10] | 13 [1 to 251]
  Met hospital discharge criteria | 1 [0 to 3] | 1 [0.8 to 3]
  Discharged from hospital | 1 [0 to 3] | 1 [0.9 to 4]
  Cleared to drive: number analyzed (Participants) | 6 | 15
  Cleared to drive | 21 [14 to 62] | 21 [15 to 71]
  Returned to work: number analyzed (Participants) | 2 | 7
  Returned to work | 9 [1 to 17] | 20 [7 to 56]
  Cessation of all opioid medications: number analyzed (Participants) | 6 | 13
  Cessation of all opioid medications | 37 [10 to 61] | 28 [6 to 336]

14. Secondary Outcome: Subject Satisfaction Survey
Description: Subjects completed a sponsor-developed survey with questions pertaining to their feelings about the treatment they received following total knee arthroplasty (TKA) surgery. Treatment Group subjects were asked to report on their experience using the SPRINT Beta Stimulation System as a method for managing post-surgical pain. Depending on the question, subjects were asked to indicate their agreement with the question (strongly disagree, agree, neutral, disagree, strongly disagree), their comfort with the therapy (very uncomfortable, a little bit uncomfortable, fairly comfortable, very comfortable), or when pain relief was felt (immediately, a few minutes later, a few hours later, more than a day later or never). Responses are presented for Treatment Group subjects for key groups of questions related to the therapy whereby answer options are considered affirmative for strongly agree/agree, very easy/easy, very comfortable/comfortable.
Time Frame: Visit 8 (4-weeks post-total knee arthroplasty (TKA))
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
Participants
  Tolerated Lead placement with some or no discomfort | 7
  Reported stimulation felt comfortable/soothing | 5
  Reported immediate pain relief (0-5 minutes) | 4
  Would recommend therapy to a friend | 7
  Would want to receive again if having another TKA | 7
  Prefer stimulation therapy to pain medication use | 7
  Wanted stimulation for longer time period before TKA surgery | 1
  Wanted stimulation for longer time period after TKA surgery | 1

15. Secondary Outcome: Number of Physical Therapy Sessions Attended Following Total Knee Arthroplasty
Description: Following discharge after total knee arthroplasty (TKA) surgery, subjects were asked to report how many physical therapy sessions they attended since the previous study visit. The median number of physical therapy sessions attended is reported for each group at each time point.
Time Frame: Visit 5 (1-week post-Total Knee Arthroplasty (TKA)), Visit 6 (2-weeks post-TKA), Visit 7 (3-weeks post-TKA), Visit 8 (4-weeks post-TKA), Visit 9 (2-months post-TKA), and Visit 10 (3-months post-TKA)
Population: Per Protocol Set - Data were not available for the following Control Group subjects: one at Visit 6, two Visit 9, and three at Visit 10.
Measure: Median (Full Range); unit: Count of visits
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 16
Count of visits
  Visit 5 (1-week Post-TKA) | 2 [1 to 3] | 2 [1 to 10]
  Visit 6 (2-weeks Post-TKA): number analyzed (Participants) | 7 | 15
  Visit 6 (2-weeks Post-TKA) | 3 [2 to 5] | 3 [2 to 14]
  Visit 7 (3-weeks Post-TKA) | 2 [1 to 3] | 3 [0 to 5]
  Visit 8 (4-weeks Post-TKA) | 2 [1 to 3] | 2 [0 to 5]
  Visit 9 (2-months Post-TKA): number analyzed (Participants) | 7 | 14
  Visit 9 (2-months Post-TKA) | 9 [4 to 12] | 5 [0 to 14]
  Visit 10 (3-months Post-TKA): number analyzed (Participants) | 7 | 13
  Visit 10 (3-months Post-TKA) | 8 [0 to 12] | 6 [0 to 12]

16. Secondary Outcome: Subject's Use of Device (Compliance)
Description: The hours of usage were recorded for each Lead (femoral and sciatic) from the SPRINT Beta stimulator throughout the study to assess the level of subject compliance with the peripheral nerve stimulation therapy. Treatment Group subjects were asked to use the device for up to 24 hrs each day. The stimulator provided the cumulative number of hours in use since the device was activated. For each timepoint for Treatment Group participants (subjects who received stimulation therapy), the median cumulative number of hours of use for each lead is presented for each timepoint.
Time Frame: Visit 4 (In-Hospital), Visit 6 (2-weeks post-Total Knee Arthroplasty (TKA)), and Visit 8 (4-weeks Post-TKA)
Population: Per Protocol Set - Treatment Group. Data were not available for the femoral or sciatic Leads for one subject at Visit 4 and two subjects at Visit 6. One subject at Visits 4, 6, 8 did not have a sciatic Lead in place.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
hours
  Visit 4 (In-Hospital): Femoral Lead: number analyzed (Participants) | 6
  Visit 4 (In-Hospital): Femoral Lead | 79 [31 to 207]
  Visit 4 (In-Hospital): Sciatic Lead: number analyzed (Participants) | 5
  Visit 4 (In-Hospital): Sciatic Lead | 73 [28 to 200]
  Visit 6 (2-weeks Post-TKA): Femoral Lead: number analyzed (Participants) | 5
  Visit 6 (2-weeks Post-TKA): Femoral Lead | 358 [190 to 519]
  Visit 6 (2-weeks Post-TKA): Sciatic Lead: number analyzed (Participants) | 4
  Visit 6 (2-weeks Post-TKA): Sciatic Lead | 373.5 [269 to 429]
  Visit 8 (4-weeks Post-TKA): Femoral Lead | 646 [266 to 744]
  Visit 8 (4-weeks Post-TKA): Sciatic Lead: number analyzed (Participants) | 6
  Visit 8 (4-weeks Post-TKA): Sciatic Lead | 633 [271 to 673]

17. Secondary Outcome: Inpatient Pain Management Experience Survey (Pain Management During Hospital Stay)
Description: Subjects completed a survey comprised of a subset of questions from the Hospital Consumer Assessment of Healthcare Providers and Systems to assess subject satisfaction with pain management during their time in the hospital for total knee arthroplasty surgery. Questions regarding experience with in-hospital pain management are reported below.
Time Frame: 1-week post-Total Knee Arthroplasty (TKA)
Population: Per Protocol Set - Data were not available for three Control Group subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 13
Participants
  During this hospital stay, how often was your pain well controlled?: Never | 0 | 0
  During this hospital stay, how often was your pain well controlled?: Sometimes | 1 | 3
  During this hospital stay, how often was your pain well controlled?: Usually | 3 | 4
  During this hospital stay, how often was your pain well controlled?: Always | 3 | 6
  During hospital stay, how often did hospital staff do everything they could to help with your pain?: Never | 0 | 0
  During hospital stay, how often did hospital staff do everything they could to help with your pain?: Sometimes | 0 | 1
  During hospital stay, how often did hospital staff do everything they could to help with your pain?: Usually | 1 | 2
  During hospital stay, how often did hospital staff do everything they could to help with your pain?: Always | 6 | 10

18. Secondary Outcome: Inpatient Pain Management Experience Survey (Pain Medicine During Hospital Stay)
Description: Subjects completed a survey comprised of a subset of questions from the Hospital Consumer Assessment of Healthcare Providers and Systems to assess subject satisfaction with pain management during their time in the hospital for total knee arthroplasty surgery. The number of subjects that responded affirmatively to the following question are reported below: "During this hospital stay, did you need medicine for pain?"
Time Frame: 1-week post-Total Knee Arthroplasty (TKA)
Population: Per Protocol - Data were not available for three Control Group subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 13
Participants | 6 | 13

19. Secondary Outcome: Inpatient Pain Management Experience Survey (Discharge Facility)
Description: Subjects completed a survey comprised of a subset of questions from the Hospital Consumer Assessment of Healthcare Providers and Systems to assess subject satisfaction with pain management during their time in the hospital for total knee arthroplasty surgery. The question regarding discharge location following hospital stay is reported below.
Time Frame: 1-week post-Total Knee Arthroplasty (TKA)
Population: Per Protocol Set - Data were not available for three Control Group subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 13
Participants
  Own home | 7 | 11
  Someone else's home | 0 | 1
  Another healthcare facility | 0 | 1

20. Secondary Outcome: Inpatient Pain Management Experience Survey (Overall Rating of Hospital)
Description: Subjects completed a survey comprised of a subset of questions from the Hospital Consumer Assessment of Healthcare Providers and Systems to assess subject satisfaction with pain management during their time in the hospital for total knee arthroplasty surgery. As part of this survey, subjects were asked to rate their hospital stay on an 11-point numerical rating scale where 0 represents "worst hospital possible" and 10 represents "best hospital possible." The median score for each group is reported.
Time Frame: 1-week post-Total Knee Arthroplasty (TKA))
Population: Per Protocol Set - Data were not available for three Control Group subjects.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 13
score on a scale | 10 [8 to 10] | 10 [7 to 10]

ADVERSE EVENTS:
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through the 12-month follow up visit. The total assessment period was approximately 13 months for each participant.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/23
Other Adverse Events (participants affected / at risk) | 12/18 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=18) | Control Group (N=23)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Not study-related
Acute Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1) — Not study-related
Pain at TKA Surgical Site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not study-related
Adverse Drug Reaction During TKA (Surgical and medical procedures) | 0 (0) | 1 (1) — Not study-related
Acute Pancreatitis and Gall Stones (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not study-related
Sepsis due to Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Not study-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment Group (N=18) | Control Group (N=23)
Skin irritation at bandage site (Skin and subcutaneous tissue disorders) | 2 (2) | 0/0 (0) — Study-Related
Skin irritation or bruising at pad and/or Lead exit site (Skin and subcutaneous tissue disorders) | 4 (4) | 0/0 (0) — Study-Related
Generalized itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
Discharge from TKA surgical incision (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
Burning sensation and swelling of knee (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
Ulcers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
Wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
New hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — One event was study-related, and the other was not
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Not Study-Related
Pain at TKA surgical site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not Study-Related
Worsening knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not Study-Related
Ankylosis of knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not Study-Related
Muscle spasming (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Study-Related
Sciatica and Piriformis Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not Study-Related
Thumb pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not Study-Related
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not Study-Related
Worsening cataract (Eye disorders) | 0 (0) | 1 (2) — Not Study-Related
Elevated blood pressure (Cardiac disorders) | 1 (1) | 0 (0) — Not Study-Related
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Not Study-Related
Bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not Study-Related
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not Study-Related
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not Study-Related
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not Study-Related
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Not Study-Related
Soreness after Lead placement (Product Issues) | 1 (1) | 0/0 (0) — Study-Related
Shocking at Lead site (Product Issues) | 1 (1) | 0/0 (0) — Study-Related
Restless Leg Syndrome flare up (Nervous system disorders) | 1 (1) | 0 (0) — Unable to determine relationship to study
Illness (General disorders) | 2 (2) | 3 (5) — Not Study-Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03286543/Prot_SAP_000.pdf